CLINICAL TRIAL: NCT03299257
Title: Donepezil for Residual Symptoms in CPAP Treated Obstructive Sleepapnea Patients: A Controlled Study
Brief Title: Donepezil, Residual Excessive Daytime Sleepiness, Obstructive Sleep Apnea
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Associação Fundo de Incentivo à Pesquisa (Other)
Responsible Party: Principal Investigator, Dalva Poyares, MD Professor, Associação Fundo de Incentivo à Pesquisa
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: RES12
Record Dates: First submitted 2017-05-11; First posted 2017-10-03 (Actual); Last update posted 2018-06-27 (Actual); Status verified 2017-09

CONDITIONS: OSA; Sleepiness
Keywords: OSA; CPAP; sleepiness; donepezil
MeSH Terms: conditions — Sleepiness

STUDY DESIGN:
Intervention Model Description: Randomized, parallel groups, 30-day trial
Who Masked: Participant, Care Provider, Investigator
Masking Description: donepezil and placebo will be dispensed to volunteers in similar pills and numbered boxes.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- donepezil treatment (Active Comparator): donepezil with 10 mg will be administered for 30 days.
  Interventions: Drug: donepezil treatment
- placebo treatment (Placebo Comparator): placebo with 10 mg placebo will be administered for 30 days.
  Interventions: Drug: donepezil treatment

INTERVENTIONS:
Drug: donepezil treatment — 30-day donepezil treatment

SUMMARY:
It is a randomized, double-blind, single-center, 30-day study. Patients aged 35-60 years, with apnea and hypopnea index and respiratory disturbance index normalized with CPAP, and Epworth Sleepiness Scale> 11. Patients undergo baseline and CPAP titration polysomnography, liquor and blood collection, Multiple Sleep Latency Test, anxiety and depression and cognitive assessments.

DETAILED DESCRIPTION:
Obstructive Sleep Apnea (OSA) is a sleep-disordered breathing characterized by recurrent episodes of total or partial obstruction of the upper airway during sleep, which can lead to cognitive, metabolic and cardiovascular consequences. More recently, OSA has been associated with worsening Alzheimer's disease symptoms. Resolving respiratory events during sleep often has a beneficial impact on these consequences. However, even after adequate and optimized treatment with continuous positive airway pressure (CPAP), about 6 to 10% of patients still remain sleepy. Given the high prevalence of OSA, this percentage represents a large number of under-treated and at-risk individuals. This residual excessive sleepiness (RES) may be related to comorbidities and cognitive alterations. Its physiopathology is still unknown. A few studies have tested modafinil as an adjunct treatment for RES patients. Since a) CPAP is ineffective in patients with RES; b) previous studies suggest some benefit with wake promoters; and c) cognitive impairment has also been reported associated with RES; the hypothesis of the present study is that donepezil improves alertness and cognition in patients with OSA and RES, evidencing the role of the cholinergic system in the pathophysiology of RES.

Objective: To evaluate the effects of donepezil on RES in adult patients treated with CPAP.

Thirty-six patients diagnosed with OSA and RES are estimated to be included. Participants will be treated with CPAP for more than 6 months with a mean use greater than 5 hours per day. After blood and cerebrospinal fluid collection, patients will be randomized into 2 groups of 30 days of treatment with donepezil or placebo. RES will be evaluated by the vigilance test and the Epworth Sleepiness Scale.

ELIGIBILITY:
Inclusion Criteria:

* Both gender, Age between 35 and 65 years;
* Confirmed diagnosis of moderate to severe OSA;
* Treatment with CPAP for at least six months;
* Persistent sleepiness with daily CPAP use compliance > 5 hours per night.

Exclusion Criteria:

* Neurological or psychiatric diseases;
* Chronic use of psychoactive drugs, other sleep disorders than OSA, visual defficiency, illiteracy.

Ages: 35 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 36 (Estimated)
Dates: Start 2018-07-06 (Estimated); Primary Completion 2018-11-04 (Estimated); Study Completion 2019-03-02 (Estimated)

PRIMARY OUTCOMES:
objective excessive daytime sleepiness | 40 days
  Maintenance Wakefulness Test
subjective excessive daytime sleepiness | 40 days
  Epworth Sleepiness Scale

SECONDARY OUTCOMES:
cognitive improvement (executive functions) | 40 days
  standard cognitive tests to evaluate executive functions

CONTACTS AND LOCATIONS:
Locations (1):
- Instituto do Sono, São Paulo, Brazil

IPD SHARING:
Plan to Share IPD: Undecided